CLINICAL TRIAL: NCT04807725
Title: Association Between IL-1 and IL-1Ra Gene Polymorphisms With Peri-implantitis
Brief Title: Analysis of Genetic Variations in Patients With Peri-implantitis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Egas Moniz - Cooperativa de Ensino Superior, CRL (Other)
Collaborators: Oral Reconstruction Foudation (Unknown)
Responsible Party: Sponsor
Other Study IDs: PHDJMC
Record Dates: First submitted 2021-03-18; First posted 2021-03-19 (Actual); Last update posted 2022-03-23 (Actual); Status verified 2022-03

CONDITIONS: Peri-Implantitis
Keywords: peri-implantitis; gene polymorphisms; interleukin-1; dental implants
MeSH Terms: conditions — Peri-Implantitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — The specimens to be retained will be cells from the oral mucosa.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Peri-implant health: Includes patients with peri implant mucosa without inflammatory signs and absence of peri-implant bone loss.
  Interventions: Genetic: Analysis of genetic polymorphisms; Other: Biochemical analysis
- Peri-implantitis: Includes patients with bleeding and / or suppuration on probing, probing depth equal or greater than 6mm and bone loss equal to or greater than 3mm.
  Interventions: Genetic: Analysis of genetic polymorphisms; Other: Biochemical analysis

INTERVENTIONS:
Genetic: Analysis of genetic polymorphisms — For the investigation of genetic polymorphisms, it will be collected a sample of cells from the jugal mucosa with the aid of a swab. The genetic analysis will be done with the DNA extraction technique followed by PCR-RFLP techniques (polymerase chain reaction followed by restriction fragment length polymorphism).
Other: Biochemical analysis — For the biochemical analysis of the inflammatory mediators IL-1beta, TNF-alpha and PGE2 a peri-implant crevicular fluid collection will be performed by inserting paper strips into peri-implant sulcus or pocket, in situations of peri-implantitis from the most affected location, while in situations of peri-implant health from the mesio-buccal location.

SUMMARY:
The primary objective of this study is to evaluate interleukin-1(IL-1) gene group polymorphisms in patients with peri-implantitis and to compare them with patients with peri-implant health (control group), taking into account smoking status, gender, age and history of periodontitis.The aim of this investigation is also to look at the levels of the inflammatory response markers IL-1 beta, prostaglandin E2 (PGE2) and tumor necrosis factor alpha (TNF alpha) in the peri-implant crevicular fluid of patients with healthy oral implants in comparison with individuals with peri-implantitis, under consideration of the patients´ individual IL-1 genotype.

The main hypothesis is that individuals carrying the polymorphism in the IL-1 gene cluster are susceptible to develop peri-implantitis through altered IL-1 and IL-1 receptor antagonist (IL-1Ra) production. A second hypothesis is that both in healthy individuals and especially pronounced in patients having peri-implantitis, an IL-1-positive genotype will result in higher levels of inflammatory cytokines (IL-1 beta, PGE2 and TNF alpha) than an IL-1- negative genotype.

Patients included in the study will be recruited from the Dental Clinic Egas Moniz implant maintenance program and will only be used for this study. All possible candidates will receive a questionnaire and if the patient's medical history is in accordance with study inclusion criteria, and if they agree to participate, informed consent will be signed. All clinical data will be collected by the same examiner.

Genes IL-1A and IL-1B control the production of the proinflammatory proteins, IL-1 alpha and IL-1 beta, respectively. IL-1RN gene controls the synthesis of the IL-1Ra, which impedes the function of IL-1alpha and IL-1beta by competing for receptor binding. Polymorphisms of the following genes will be analyzed: IL-1A-889, IL-1B + 3954, IL-1B-511 and IL-1 RN from patients with peri-implantitis and peri-implant health. For the investigation of genetic polymorphisms, it will be collected a sample of cells from the jugal mucosa with the aid of a swab.

For the biochemical analysis of the inflammatory mediators IL-1 beta, TNF alpha and PGE2 a peri-implant crevicular fluid collection will be performed by inserting paper strips into peri-implant sulcus or pocket, in situations of peri-implantitis from the most affected location, while in situations of peri-implant health from the mesio-buccal location.

DETAILED DESCRIPTION:
The study will be conducted according to the principles of the Helsinki Declaration (reviewed in 2013). Appropriate measures will be taken for the protection of patient data. The study was approved by Instituto Universitário Egas Moniz (IUEM) Scientific Council on 3 July 2019 and the approval of the Ethics Committee of Egas Moniz was received on 24 July 2019. Authorization was also obtained by the Clinical Direction of Egas Moniz Dental Clinic to carry out research work at the Clinic of the University.

The study will consist of two groups, the first consisting of patients with peri-implantitis (bleeding and / or suppuration on probing, probing depth (PD) equal or greater than 6mm and bone loss equal to or greater than 3mm) and the second group (control group) formed by patients with peri-implant health (peri implant mucosa without inflammatory signs and absence of peri-implant bone loss). The definition of peri-implantitis and peri-implant health will be in accordance with the new classification of periodontal and peri-implant diseases (American Academy of Periodontology (AAP) and European Federation of Periodontology (EFP) 2017)

A peri-implant probing examination (6 locations with a CP12 graduated periodontal probe) and evaluation of plaque accumulation and gingival indexes (4 locations) will be performed as usual at implant maintenance appointments. The presence of bleeding on probing or pus will also be evaluated. An implant control radiograph will be taken in cases where there is a probing depth more than 6mm. All clinical data will be collected by the same examiner. Prior to the study, a training and calibration exercise will be performed for PD measurements using patients not included in the study.

The periodontal condition of the patients will be also evaluated. To consider periodontal health, patients should have the following clinical characteristics: up to 10% of locations with bleeding on probing, absence of erythema and edema, absence of patient symptoms, absence of clinical attachment loss and bone loss and PD < 3mm (AAP and EFP 2017). A patient is a periodontitis case if: interdental clinical attachment loss is detectable at least 2 non-adjacent teeth, or buccal or oral clinical attachment loss >3mm with pocketing >3mm is detectable at least 2 teeth. The classification of periodontitis will be done on a multi-dimensional staging and grading system.

In the case of a peri-implant health situation, plaque control measures will be taken, while in cases of peri-implantitis the patient will be referred for a specific treatment appointment. In situations of patients with more than one implant affected by peri-implantitis, the one with the greatest bone loss will be chosen for the study.

The genetic analysis will be done at the IUEM Molecular Biology Laboratory with the DNA extraction technique followed by polymerase chain reaction followed by restriction fragment length polymorphism.

For the biochemical analysis the paper strips will be inserted into the peri-implant sulcus/ pocket until resistance is felt, waiting 30 seconds before removal. Visually contaminated samples (blood) will be discarded. Subsequently paper strips will be placed on Periotron® 8000 (Periotron Ide-interstate, NY, USA) for quantification of the collected peri-implant crevicular fluid volume. The strips of paper will then be placed in eppendorf tubes with filter and frozen at -80ºC until shipment to the Universidad Complutense de Madrid. At this university, the concentration of inflammatory mediators IL-1 beta and TNF alpha will be analyzed using multiplexed fluorescent sphere immunoassays using the Luminex® 100/200™ system and PGE2 by enzyme-linked immunosorbent assay (ELISA).

The prevalence of IL-1 gene group polymorphisms in patients with peri-implantitis and healthy ones will be compared by using appropriate inferential statistics methodologies (bivariate analysis/association tests), taking into account several sociodemographic and clinical variables: smoking status, gender, age and history of periodontitis. Based on a medium effect size (w=0.3), with 80% power and a 5% alpha level, the sample size for this study was calculated as n=88, thus, n= 44 for each group (periimplantitis and peri-implant health). Further, a multivariable regression logistic model will be constructed in order to evaluate the effect of those covariables and quantify the risk, through determination of the correspondent adjusted Odds Ratio (OR), towards the presence of peri-implantitis. Additionally, the levels of the inflammatory response markers IL-1 beta, PGE2 and TNF-alpha, present in the peri-implant crevicular fluid, will be compared between the group of patients with peri-implantitis and the patients with healthy oral implants, taking into account the above mentioned variables, by using appropriate inferential statistics methodologies (parametric/non parametric tests). All inferential analysis will be performed at a 5% significance level.

ELIGIBILITY:
Inclusion Criteria:

* patients with Caucasian parents and grandparents
* patients with dental implants placed at the Dental Clinic Egas Moniz or out
* patients with peri-implantitis diagnosis
* implants in function for at least 1 year
* patients included in a periodontal / peri-implant support program
* patients who agree to participate in the study and sign informed consent

Exclusion Criteria:

* patients with any systemic condition that affects the immune system
* pregnant women
* patients who have taken chronic antibiotics or anti-inflammatory drugs in the last 6 months
* patients who have undergone peri-implant treatment in the area to be evaluated

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients included in the study will be recruited from the Dental Clinic Egas Moniz implant maintenance program and will only be used for this study. All possible candidates will receive a questionnaire and if the patient's medical history is in accordance with study inclusion criteria, and if they agree to participate, informed consent will be signed.
Sampling Method: Non-Probability Sample
Enrollment: 88 (Estimated)
Dates: Start 2021-03-09 (Actual); Primary Completion 2022-07-29 (Estimated); Study Completion 2022-07-29 (Estimated)

PRIMARY OUTCOMES:
Frequency of Participants with polymorphism in the IL-1 gene cluster | 1 month after sample collection
  In the IL-1A-889 gene, two possible alleles are expected to be found, allele 1 (83 base pairs (bp) + 16 bp), allele 2 - allele with nucleotide sequence changed (99 bp). In the IL-1B + 3954 gene, two possible alleles are expected to be found, allele 1 (12 bp + 85 bp + 97 bp), allele 2 (12 bp + 182 bp). In the IL-1B-511 gene, two possible alleles are expected to be found, allele 1 (190bp + 114bp), allele 2 (304 bp). In relation to the polymorphism of the IL-1RN gene, 5 possible alleles are expected to be found according to the repeated base pair sequences: allele 1 (410 bp), allele 2 (240 bp), allele 3 (500 bp), allele 4 (325 bp), allele 5 (595 bp).

SECONDARY OUTCOMES:
Concentration of inflammatory response markers IL-1 beta, PGE2 and TNF-alpha | 1 month after sample collection
  The paper strips with peri-implant crevicular fluid (PICF) will be placed on Periotron® 8000 (Periotron Ide-interstate, NY, USA) for quantification of the collected PICF volume.The concentration of inflammatory mediators IL-1beta and TNF-alpha will be analyzed using multiplexed fluorescent sphere immunoassays using the Luminex® 100/200™ system and PGE2 by ELISA (enzyme-linked immunosorbent assay).

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo Alves, Phd, Principal Investigator — Egas Moniz
Locations (1):
- Instituto Universitário Egas Moniz, Almada, Monte de Caparica, Portugal

IPD SHARING:
Plan to Share IPD: No
The collections of DNA samples were collected only for the purpose of analyzing the polymorphisms of the IL-1 gene group. Participants authorized their collection only for this purpose. For ethical and confidentiality reasons, these samples may not be accessible to other researchers. DNA samples will be eliminated after conducting the study.

REFERENCES:
- [Background] Chen X, Zhao Y. Genetic Involvement in Dental Implant Failure: Association With Polymorphisms of Genes Modulating Inflammatory Responses and Bone Metabolism. J Oral Implantol. 2019 Aug;45(4):318-326. doi: 10.1563/aaid-joi-D-18-00212. Epub 2019 Jun 17. PMID 31207194
- [Background] Duarte PM, de Mendonca AC, Maximo MB, Santos VR, Bastos MF, Nociti Junior FH. Differential cytokine expressions affect the severity of peri-implant disease. Clin Oral Implants Res. 2009 May;20(5):514-20. doi: 10.1111/j.1600-0501.2008.01680.x. Epub 2009 Mar 11. PMID 19302394
- [Background] Feloutzis A, Lang NP, Tonetti MS, Burgin W, Bragger U, Buser D, Duff GW, Kornman KS. IL-1 gene polymorphism and smoking as risk factors for peri-implant bone loss in a well-maintained population. Clin Oral Implants Res. 2003 Feb;14(1):10-7. doi: 10.1034/j.1600-0501.2003.140102.x. PMID 12562360
- [Background] Gruica B, Wang HY, Lang NP, Buser D. Impact of IL-1 genotype and smoking status on the prognosis of osseointegrated implants. Clin Oral Implants Res. 2004 Aug;15(4):393-400. doi: 10.1111/j.1600-0501.2004.01026.x. PMID 15248873
- [Background] Lachmann S, Kimmerle-Muller E, Axmann D, Scheideler L, Weber H, Haas R. Associations between peri-implant crevicular fluid volume, concentrations of crevicular inflammatory mediators, and composite IL-1A -889 and IL-1B +3954 genotype. A cross-sectional study on implant recall patients with and without clinical signs of peri-implantitis. Clin Oral Implants Res. 2007 Apr;18(2):212-23. doi: 10.1111/j.1600-0501.2006.01322.x. PMID 17348886
- [Background] Petkovic-Curcin A, Zeljic K, Cikota-Aleksic B, Dakovic D, Tatic Z, Magic Z. Association of Cytokine Gene Polymorphism with Peri-implantitis Risk. Int J Oral Maxillofac Implants. 2017 Sep/Oct;32(5):e241-e248. doi: 10.11607/jomi.5814. PMID 28906511
- [Background] He K, Jian F, He T, Tang H, Huang B, Wei N. Analysis of the association of TNF-alpha, IL-1A, and IL-1B polymorphisms with peri-implantitis in a Chinese non-smoking population. Clin Oral Investig. 2020 Feb;24(2):693-699. doi: 10.1007/s00784-019-02968-z. Epub 2019 May 24. PMID 31127430
- [Background] McDowell TL, Symons JA, Ploski R, Forre O, Duff GW. A genetic association between juvenile rheumatoid arthritis and a novel interleukin-1 alpha polymorphism. Arthritis Rheum. 1995 Feb;38(2):221-8. doi: 10.1002/art.1780380210. PMID 7848312
- [Background] Tarlow JK, Blakemore AI, Lennard A, Solari R, Hughes HN, Steinkasserer A, Duff GW. Polymorphism in human IL-1 receptor antagonist gene intron 2 is caused by variable numbers of an 86-bp tandem repeat. Hum Genet. 1993 May;91(4):403-4. doi: 10.1007/BF00217368. PMID 8500797
- [Background] Hamdy AA, Ebrahem MA. The effect of interleukin-1 allele 2 genotype (IL-1a(-889) and IL-1b(+3954)) on the individual's susceptibility to peri-implantitis: case-control study. J Oral Implantol. 2011 Jun;37(3):325-34. doi: 10.1563/AAID-JOI-D-09-00117.1. Epub 2010 Jun 16. PMID 20594066
- [Background] Dereka X, Mardas N, Chin S, Petrie A, Donos N. A systematic review on the association between genetic predisposition and dental implant biological complications. Clin Oral Implants Res. 2012 Jul;23(7):775-88. doi: 10.1111/j.1600-0501.2011.02329.x. Epub 2011 Dec 12. PMID 22151432
- [Background] Laine ML, Leonhardt A, Roos-Jansaker AM, Pena AS, van Winkelhoff AJ, Winkel EG, Renvert S. IL-1RN gene polymorphism is associated with peri-implantitis. Clin Oral Implants Res. 2006 Aug;17(4):380-5. doi: 10.1111/j.1600-0501.2006.01249.x. PMID 16907768
- [Background] Huynh-Ba G, Lang NP, Tonetti MS, Zwahlen M, Salvi GE. Association of the composite IL-1 genotype with peri-implantitis: a systematic review. Clin Oral Implants Res. 2008 Nov;19(11):1154-62. doi: 10.1111/j.1600-0501.2008.01596.x. PMID 18983319
- [Background] Andreiotelli M, Koutayas SO, Madianos PN, Strub JR. Relationship between interleukin-1 genotype and peri-implantitis: a literature review. Quintessence Int. 2008 Apr;39(4):289-98. PMID 19081897
- [Background] Liao J, Li C, Wang Y, Ten M, Sun X, Tian A, Zhang Q, Liang X. Meta-analysis of the association between common interleukin-1 polymorphisms and dental implant failure. Mol Biol Rep. 2014 May;41(5):2789-98. doi: 10.1007/s11033-014-3133-6. Epub 2014 Jan 23. PMID 24452718
- [Background] Fourmousis I, Vlachos M. Genetic Risk Factors for the Development of Periimplantitis. Implant Dent. 2019 Apr;28(2):103-114. doi: 10.1097/ID.0000000000000874. PMID 30865053
- [Background] Vaz P, Gallas MM, Braga AC, Sampaio-Fernandes JC, Felino A, Tavares P. IL1 gene polymorphisms and unsuccessful dental implants. Clin Oral Implants Res. 2012 Dec;23(12):1404-13. doi: 10.1111/j.1600-0501.2011.02322.x. Epub 2011 Nov 10. PMID 22092925